CLINICAL TRIAL: NCT00455390
Title: Evaluation of the Effects of Post-Immediate Psychotherapeutic Interventions in Secondary Prevention of Psychotraumatic Disorders
Acronym: IPPI A
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Groupe Francais d'Epidemiologie Psychiatrique (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IPPI A
Record Dates: First submitted 2007-04-02; First posted 2007-04-03 (Estimated); Last update posted 2007-04-03 (Estimated); Status verified 2007-04

CONDITIONS: PTSD Post Traumatic Syndrome Disorder
Keywords: Post immediate Psychotherapeutic Intervention; Psychotraumatic disorders; PTSD post traumatic syndrome disorder; CUMP Cellules d'Urgence Médico Psychologique

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Post-immediate Psychotherapeutic Intervention

SUMMARY:
Argumentation The frequency of post-traumatic syndrome disorder (PTSD) is estimated around 1% of the entire European population. In some specific populations, this percentage increases (soldiers - 15 to 22%, war or persecuted refugees - 80%, post office or bank employees submitted to an hold-up - 17%, firemen - 10 to 30%, emergency care employees - 11%, people who underwent a terrorist attack or any violence - 20 to 65%...)

Prevention is yet poor, secondary prevention trying to avoid a post traumatic disorder apparition early after the traumatic event. There is currently two types of secondary prevention :

* Mitchell's debriefing based upon stress and its theories, using cognitive and behavioural approaches
* French debriefing (post-immediate psychotherapeutic intervention) based on the traumatism, never realised before second day post event and applied by mental health professionals.

The current controversy of the Mitchell's debriefing leads us to evaluate the post-immediate psychotherapeutic intervention, never evaluated yet.

Scientific Objectives Primary objective: To verify that post-immediate psychotherapeutic interventions (proposed after 2 days and before the end of first month post event) decrease incidence, duration and intensity of psychotraumatic disorders at one year, versus a control group.

Secondary objectives :

* To document the efficacy of these interventions regarding professional, social and familial adaptation.
* To identify predictive factors of response to this strategy.

Method Experimental Design National multicentered, randomized, single blind study Study Population 330 men or women aged 18 to 65, subjected to a potentially traumatic event (criteria A1, DSM IV) and having presented an emotional reaction (intense fear, impotency or horror, criteria A2, DSM IV). This event must have happened within 8 days prior randomization. Patients treated with βblockers and patients suffering from psychopathologic disorders won't be considered for the study.

Outcome measures Primary outcome: PTSD frequency (on the basis of questionnaire CAPS).

Secondary outcome:

* Complete and subsyndormic PTSD occurence (CAPS),
* Intensity of psychotraumatic disorders (Sheehan scale),
* Psychopathologic disorder frequency (CIDI SF),
* Evolution of anxiety/depression (HAD scale),
* Alcoholization frequency (CAGE scale),
* Frequency of somatic adverse events,
* Access to health care (number and types of contacts).

Expected benefits The post-immediate psychotherapeutic intervention shall avoid psychological disorders apparition or improve its symptoms. This would decrease consequences on personal life (social, relational and professional).

The study results will allow a better knowledge of these post traumatic disorders.

DETAILED DESCRIPTION:
Intervention:

Group 1: Post-immediate psychotherapeutic intervention, 2 to 3 seances within the first month following the potentially traumatic event. Each intervention last about 45 minutes.

Group 2-control: no psychotherapeutic intervention, only 2 to 3 supporting sessions.

Eligibility criteria:

Inclusion criteria

* men or women aged 18 to 65,
* subjected to a potentially traumatic event (criteria A1, DSM IV),
* having presented an emotional reaction (intense fear, impotency or horror, criteria A2, DSM IV),
* potentially traumatic event happening within 8 days prior randomization.

Non inclusion criteria

* patients treated with βblockers ,
* patients suffering from psychopathologic disorders within 15 days prior randomization (Axe I DSM IV),
* physical injuries avoiding patient's participation to the study,
* hospitalization > 72 hours post event,
* traumatic event related to a process of victimisation (domestic violences),
* no informed consent signed

Study type:

Randomized, single blind trial on two parallel groups. Randomization stratified on sex and human design.

Number of patients:

330 in 18 clinical centres

ELIGIBILITY:
Inclusion Criteria:

* men or women aged 18 to 65,
* subjected to a potentially traumatic event (criteria A1, DSM IV),
* having presented an emotional reaction (intense fear, impotency or horror, criteria A2, DSM IV),
* potentially traumatic event happening within 8 days prior randomization.

Exclusion Criteria:

* patients treated with βblockers ,
* patients suffering from psychopathologic disorders within 15 days prior randomization (Axe I DSM IV),
* physical injuries avoiding patient's participation to the study,
* hospitalization > 72 hours post event,
* traumatic event related to a process of victimisation (domestic violences),
* no informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330
Dates: Start 2007-01; Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
PTSD frequency (questionnaire CAPS at 1, 3, 6 and 12 months )

SECONDARY OUTCOMES:
Complete and subsyndormic PTSD occurence (CAPS at 1, 3, 6 and 12 months)
Intensity of psychotraumatic disorders (Sheehan scale at 1, 3, 6 and 12 months).
Psychopathologic disorder frequency (CIDI SF at baseline and at 1, 3, 6 and 12 months).
Evolution of anxiety/depression (HAD scale after first therapy session and at 1, 3, 6 and 12 months).
Alcoholization frequency (CAGE scale at baseline and at 1, 3, 6 and 12 months).
Frequency of somatic adverse events (at each visit).
Access to health care (number and types of contacts, at each visit).

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie PRIETO, MDH, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Edouard Herriot - SAMU, Lyon, Auvergne-Rhône-Alpes, France